CLINICAL TRIAL: NCT01759056
Title: A Multicenter, Double-Blind, Placebo-Controlled, Ascending-Dose, Repeat-Dose Safety and Pharmacokinetic Investigation of a Delayed-Release, Enteric-Coated Capsule Formulation of AVX 470 [Anti-TNF (Tumor Necrosis Factor) Globulin (Bovine)] in Patients With Active Ulcerative Colitis
Brief Title: Evaluation of an Oral Anti-TNF Antibody in Patients With Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avaxia Biologics, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB1101; 2012-004850-27 (EudraCT Number)
Record Dates: First submitted 2012-12-24; First posted 2013-01-02 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVX 470 (Active Comparator): AVX 470 0.2 g(Cohort 1), 1.6 g (Cohort 2) and 3.5 g (Cohort 3) will be administered daily for 28 days
  Interventions: Drug: AVX 470
- Placebo (Placebo Comparator): Placebo will be administered daily for 28 days as a comparator with AVX-470 (all dose groups)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVX 470 — active comparator
  Arms: AVX 470
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability as well as the pharmacodynamic effects of multiple doses of AVX-470 administered orally in patients with active ulcerative colitis.

DETAILED DESCRIPTION:
There is a significant unmet medical need for effective oral pharmacologic therapies for inflammatory bowel diseases such as ulcerative colitis. Current anti-TNF therapies, including infliximab and adalimumab, are effective treatments for these conditions, but they must be administered by intravenous or subcutaneous injection. The major safety concerns associated with the use of injectable anti-TNF therapies are infection, demyelinating disease, and lymphoma, all of which are the result of systemic exposure. These uncommon but serious side effects have limited the use of systemic anti-TNF antibody therapy to patients with severe disease that have failed to respond to first-line treatments.

AVX-470 is purified immunoglobulin (Ig) from the colostrum (early milk) of cows immunized with recombinant human tumor necrosis factor (rhTNF). AVX-470 is formulated in delayed-release enteric-coated capsules designed to protect the capsule contents from gastric acids following oral administration and to provide localized delivery to sites of inflammation in the distal intestine. Prior clinical experience with bovine Ig therapies in other human diseases suggests that AVX-470 will not be absorbed to any significant extent, meaning that systemic exposure could be minimized. The development of oral anti-TNF therapy targeting local intestinal disease activity might reduce the risks associated with injectable anti-TNF therapy and allow the convenience of oral dosing.

The present study is a first-in-human, Phase 1 clinical study. It is primarily intended to evaluate the safety and tolerability of multiple doses of AVX-470 administered orally to patients with active ulcerative colitis.

Animal models of ulcerative colitis using a mouse-specific TNF antibody derived from bovine colostrum demonstrated a 50% or more reduction in tissue TNF, TNF-messenger ribonucleic acid (mRNA), interleukin (IL)-6 mRNA, and myeloperoxidase and lowering of colonic inflammatory activity. Twenty-eight-day toxicology studies demonstrated no clinical or histologic findings in exposures above the intended clinical dose range.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 75, inclusive
* Established diagnosis of ulcerative colitis involving the sigmoid colon or proximal segments of bowel
* Total Mayo score between 5-12, inclusive, with endoscopic subscore of the Mayo score ≥ 2 and > 15 cm of involvement beyond the anal verge

Exclusion Criteria:

* Women with a positive pregnancy test, who are breastfeeding, or who intend to become pregnant during the course of the study
* Diagnosis of Crohn's disease, microscopic colitis or indeterminate colitis
* Presence of ileostomy or colostomy, or history of prior colon resection
* Patients with planned hospitalization or surgery during the course of the study
* Known allergy to milk proteins, red meat or cornstarch
* Stools positive for enteric infection, including parasitic, or C. difficile toxin within 28 days of screening
* Documented presence of Hetatitis B (HBsAg), Hepatitis C (HCV), or HIV
* Presence of dysplasia of any grade on colonoscopic biopsies
* Treatment for cancer (excluding non-melanomatous cancer of the skin or cervical carcinoma in situ) or lymphoproliferative disorder (including lymphoma) within 5 years
* History of tuberculosis (TB) or Listeria infection, or known exposure to another person with active TB disease within 12 weeks of screening; or history of past or current infection with different opportunistic infections
* History of TNF inhibitor (infliximab, adalimumab or certolizumab pegol) use with primary treatment failure. Secondary treatment failures due to intolerance, allergic reaction, or loss of response will not constitute a basis for exclusion. Oral immunosuppressives, mesalamine, and corticosteroids (up to 20mg of prednisone per day) will be permitted so long as these medications are stable for defined periods of time before study participation commences.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AVX-470 over 28 days of treatment | 5 weeks
  Assessments weekly during treatment and 1 week post treatment

SECONDARY OUTCOMES:
Pharmacokinetics (serum, stool and gastrointestinal mucosal tissue levels) of AVX-470 | 4 weeks
Measure the induction of or change in a human anti-bovine immunoglobulin antibody (HABA) response to AVX 470 | 4 weeks

OTHER OUTCOMES:
Clinical response to AVX 470 in ulcerative colitis, as assessed by the total Mayo score and subscores, after 28 days of treatment compared to Baseline | 4 weeks
Effect of AVX 470 on endoscopic healing in ulcerative colitis, as assessed by the endoscopic subscore of the total Mayo score and the Ulcerative Colitis Index of Severity (UCEIS), after 28 days of treatment compared to Baseline | 4 weeks
Evaluate the effects of AVX 470 on biomarkers of ulcerative colitis activity over 28 days of treatment compared to Baseline | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott Harris, MD, Study Director — Avaxia Biologics, Incorporated
Locations (16):
- United States (9):
  - Anaheim Clinical Trials, Anaheim, California
  - Rocky Mountain Gastroenterology Associates, Lakewood, Colorado
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Center for Digestive and Liver Disease, Mexico, Missouri
  - Remington-Davis, Inc., Columbus, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Nashville Medical Research Institute, Nashville, Tennessee
- Belgium (2):
  - Gastro-Enterologie, Ghent
  - Gastro-enterologie, Leuven
- Canada (2):
  - The Northern Alberta Clinical Trials and Research Centre, Edmonton, Alberta
  - Toronto Digestive Disease Associates, Toronto, Ontario
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Debrecen
  - Kenézy Kórház Rendelöintézet Egészségügyi Szolgáltató Kft., Debrecen

REFERENCES:
- [Derived] Harris MS, Hartman D, Lemos BR, Erlich EC, Spence S, Kennedy S, Ptak T, Pruitt R, Vermeire S, Fox BS. AVX-470, an Orally Delivered Anti-Tumour Necrosis Factor Antibody for Treatment of Active Ulcerative Colitis: Results of a First-in-Human Trial. J Crohns Colitis. 2016 Jun;10(6):631-40. doi: 10.1093/ecco-jcc/jjw036. Epub 2016 Jan 28. PMID 26822613
- [Derived] Hartman DS, Tracey DE, Lemos BR, Erlich EC, Burton RE, Keane DM, Patel R, Kim S, Bhol KC, Harris MS, Fox BS. Effects of AVX-470, an Oral, Locally Acting Anti-Tumour Necrosis Factor Antibody, on Tissue Biomarkers in Patients with Active Ulcerative Colitis. J Crohns Colitis. 2016 Jun;10(6):641-9. doi: 10.1093/ecco-jcc/jjw026. Epub 2016 Jan 22. PMID 26802087